CLINICAL TRIAL: NCT03424018
Title: A Phase 3, Open-Label Long-Term Extension Study to Evaluate the Safety and Efficacy of BMN 111 in Children With Achondroplasia
Brief Title: An Extension Study to Evaluate the Efficacy and Safety of BMN 111 in Children With Achondroplasia
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 111-302; 2017-002404-28 (EudraCT Number)
Record Dates: First submitted 2017-12-28; First posted 2018-02-06 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: Achondroplasia
Keywords: ACH; Achondroplasia; Bone Diseases; Bone Diseases, Developmental; Dwarfism; Genetic Diseases, Inborn; Musculoskeletal Diseases; Natriuretic Agents; Natriuretic Peptide, C-Type; Osteochondrodysplasias; Physiological Effects of Drugs; Skeletal Dysplasias
MeSH Terms: conditions — Achondroplasia; Bone Diseases; Bone Diseases, Developmental; Dwarfism; Genetic Diseases, Inborn; Musculoskeletal Diseases; Osteochondrodysplasias | interventions — vosoritide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BMN 111 (Experimental)
  Interventions: Drug: BMN 111

INTERVENTIONS:
Drug: BMN 111 — Subcutaneous injection of recommended dose of BMN 111 based on weight-band dosing once daily.
  Other Names: Vosoritide; Modified recombinant human C-type natriuretic peptide

SUMMARY:
The intent and design of this Phase 3 study is to assess BMN 111 as a therapeutic option for the treatment of children with Achondroplasia

ELIGIBILITY:
Inclusion Criteria:

* Must have completed Study 111-301
* Female >= 10 years old or who have begun menses must have a negative pregnancy test at the Baseline Visit and be willing to have additional pregnancy tests during the study
* If sexually active, willing to use a highly effective method of contraception while participating in the study
* Are willing and able to perform all study procedures
* Parent(s) or guardian(s) are willing and able to provide written, signed informed consent after the nature of the study has been explained and prior to performance of any research-related procedure. Also, subjects under the age of majority are willing and able to provide written assent (if required by local regulations or the IRB/IEC) after the nature of the study has been explained and prior to performance of any research-related procedure. Subjects who reach the age of majority in their country while the study is ongoing will be asked to provide their own written consent again upon reaching the legal age of majority.

Exclusion Criteria:

* Permanently discontinued BMN 111 or placebo prior to completion of the 111-301 study
* Have a clinically significant finding or arrhythmia on Baseline ECG that indicates abnormal cardiac function
* Evidence of decreased growth velocity (<1.5 cm/year) as assessed over a period of at least 6 months or of growth plate closure (proximal tibia, distal femur) through bilateral lower extremity X-rays.
* Require any investigational agent prior to completion of study period
* Current therapy with medications known to alter renal function
* Pregnant or breastfeeding or plan to become pregnant during study
* Concurrent disease or condition that, in the view of the investigator, would interfere with study participation or safety evaluations, for any reason.
* Have a condition or circumstance that, in the view of the investigator, places the subject at high risk for poor treatment compliance or for not completing the study.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2031-06 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Change from baselines in mean annualized growth velocity | Through study completion, an average of 1 year
  Long term efficacy as measured by change in annualized growth velocity

SECONDARY OUTCOMES:
Changes in health-related quality of life as measured by the Quality of Life in Short-Statured Youth questionnaire | Through study completion, every 6-12 months
Potential changes in daily activity performance as measured by Activities of Daily Living questionnaire | Through study completion, every 12 months
Characterize maximum concentration (Cmax) of BMN 111 in plasma | Through study completion, every 12 months
Characterize the area under the plasma concentration time-curve from time 0 to infinity (AUC0-∞) | Through study completion, every 12 months
Characterize the area under the plasma concentration time-curve from time 0 to the last measurable concentration (AUC0-t) | Through study completion, every 12 months
Characterize the elimination half-life of BMN 111 (t1⁄2) | Through study completion, every 12 months
Characterize the apparent clearance of drug | Through study completion, every 12 months
Characterize the apparent volume of distribution based upon the terminal phase (Vz/F) | Through study completion, every 12 months
Characterize the amount of time BMN 111 is present at maximum concentration (Tmax) | Through study completion, every 12 months
BMN 111 Activity Biomarkers | Through study completion, every 12 months
  BMN 111 activity will be assessed by measuring bone and collagen metabolism
Evaluate change from baseline in body proportion ratios of the extremities | Through study completion, every 6 months
Effect of BMN 111 on bone morphology and quality | Through study completion, every 12 months for DXA or 2 years for X-ray
  The effect of BMN 111 on bone morphology/quality will be assessed by measuring bone mineral density via X-Ray and Dual X-ray Absorptiometry
Final Adult Height | Up to at least 16 years of age for females and 18 years of age for males
  Height at 16 years for females and 18 years for males

OTHER OUTCOMES:
Optional exploratory genomic biomarker analysis | Once through study completion
  Exploratory genomic analysis of genes associated with CNP signaling

CONTACTS AND LOCATIONS:
Locations (24):
- United States (11):
  - Children's Hospital & Research Center Oakland, Oakland, California
  - Harbor - UCLA Medical Center, Torrance, California
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Emory University, Atlanta, Georgia
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - University of Missouri, Columbia, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Baylor College of Medicine, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Medical College of Wisconsin, Children's Hospital, Milwaukee, Wisconsin
- Australia (2):
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Murdoch Children's Research Institute, Parkville, Victoria
- Germany (2):
  - Otto-von-Gericke Universitaet, Universitaetskinderklinik, Magdeburg
  - Universitätsklinikum Münster, Münster
- Japan (3):
  - Osaka University Hospital, Osaka
  - Saitama Children's Medical Center, Saitama
  - Tokushima University Hospital, Tokushima
- Spain (3):
  - Institut Catala de Traumatologica I Medicina de l'Esport, Barcelona
  - Hospital Sant Joan de Deu, Barcelona
  - Hospital Universitario Virgen de la Victoria, Málaga
- Acibadem University School of Medicine, Istanbul, Turkey (Türkiye)
- United Kingdom (2):
  - Guy's and St. Thomas NHS Foundation Trust Evelina Children's Hospital, London
  - Sheffield Children's NHS Foundation Trust, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Savarirayan R, Irving M, Wilcox WR, Bacino CA, Hoover-Fong JE, Harmatz P, Polgreen LE, Palm K, Prada CE, Kubota T, Arundel P, Kotani Y, Leiva-Gea A, Bober MB, Hecht JT, Legare JM, Lawrinson S, Low A, Sabir I, Huntsman-Labed A, Day JRS. Sustained growth-promoting effects of vosoritide in children with achondroplasia from an ongoing phase 3 extension study. Med. 2025 May 9;6(5):100566. doi: 10.1016/j.medj.2024.11.019. Epub 2024 Dec 30. PMID 39740666
- [Derived] Qi Y, Chan ML, Mould DR, Larimore K, Fisheleva E, Cherukuri A, Day J, Savarirayan R, Irving M, Bacino CA, Hoover-Fong J, Ozono K, Mohnike K, Wilcox WR, Bober MB, Henshaw J. Development of a Weight-Band Dosing Approach for Vosoritide in Children with Achondroplasia Using a Population Pharmacokinetic Model. Clin Pharmacokinet. 2024 May;63(5):707-719. doi: 10.1007/s40262-024-01371-6. Epub 2024 Apr 23. PMID 38649657
- See also: NIH Genetics Home Reference related topics: Achondroplasia — https://ghr.nlm.nih.gov/condition/achondroplasia
- See also: Description NIH Genetic and Rare Diseases Information Center resources: Achondroplasia — https://rarediseases.info.nih.gov/diseases/8173/achondroplasia
- See also: U.S. FDA Resources — https://clinicaltrials.gov/ct2/info/fdalinks